CLINICAL TRIAL: NCT00004076
Title: A Phase I Study to Evaluate MAG-CPT (PNU 166148) Given as One Single Intravenous Administration Every 4 Weeks in Patients With Advanced Solid Tumors
Brief Title: PNU 166148 in Treating Patients With Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Glasgow (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067285; CRC-BOC-98OMCP001; EU-99009; P-UPJOHN-98OMCP001
Record Dates: First submitted 1999-12-10; First posted 2004-06-17 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2000-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Drug: mureletecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of PNU 166148 in treating patients who have metastatic solid tumors that have not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety profile, maximum tolerated dose, and dose limiting toxicities of PNU 166148 in patients with metastatic, refractory solid tumors. II. Define a recommended dose of PNU 166148 for a Phase II study. III. Determine the pharmacokinetic profile and molecular weight distribution of PNU 166148 and the pharmacokinetic profile of free camptothecin in these patients. IV. Assess any evidence of antitumor activity in these patients treated with this regimen.

OUTLINE: This is a dose escalation, open label, multicenter study. Patients receive PNU 166148 IV over 30 minutes. Treatment repeats every 4 weeks for 3-6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of PNU 166148 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 3-6 patients experience dose limiting toxicity. Patients are followed for 30 days, and then monthly thereafter only for resolution of adverse events that occurred while on study and were attributable to study drug, unless another antitumor treatment is begun.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic, refractory solid tumors for which no curative therapy exists No more than 2 prior chemotherapy regimens for metastatic disease No prior high dose chemotherapy regimen requiring bone marrow transplantation or peripheral blood stem cell transplantation No hematologic malignancies No brain or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal (no greater than 1.5 times upper limit of normal (ULN) if liver metastases present) SGOT and SGPT normal (no greater than 5 times ULN if liver metastases present) Hepatitis B negative Renal: Creatinine less than 1.5 mg/dL EDTA clearance greater than 60 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception during and for 6 months after study No severe concurrent nonmalignant disease that would preclude protocol therapy HIV negative No AIDS related illness No mental incapacity

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 4 weeks since prior immunotherapy and recovered No concurrent biological response modifier therapy or immunotherapy No concurrent prophylactic growth factors Chemotherapy: See Disease Characteristics No prior camptothecins (e.g., irinotecan or topotecan) At least 4 weeks since other prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered No other concurrent chemotherapy Endocrine therapy: At least 4 weeks since prior hormonal therapy and recovered No concurrent corticosteroids used as anticancer therapy No other concurrent hormonal therapy Radiotherapy: No prior radiotherapy to greater than 25% of bone marrow At least 4 weeks since other prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified Other: No concurrent investigational drug or participation in other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-06

CONTACTS AND LOCATIONS:
Overall Officials: Chris Twelves, MD, BMedSci, FRCP, Study Chair — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland